CLINICAL TRIAL: NCT02216279
Title: Phase-II Study of the Use of PulmoBind for Molecular Imaging of Pulmonary Hypertension
Acronym: PB-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PulmoBind II safety Trial
Record Dates: First submitted 2014-06-27; First posted 2014-08-13 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary; Hypertension; PH; PulmoBind; Imaging
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension | interventions — adrenomedullin (22-52), glycyl-glycyl-alanyl-glycyl-cysteinyl-(PEG)4-cysteinyl-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary Hypertension Patients (Experimental): PulmoBind is a peptide derived from human adrenomedullin (hAM1-52), labelled with 99mTc (imaging isotope used in clinical medicine).
  Interventions: Drug: PulmoBind
- Control Non-Smoking Participants (Active Comparator): PulmoBind is a peptide derived from human adrenomedullin (hAM1-52), labelled with 99mTc (imaging isotope used in clinical medicine).
  Interventions: Drug: PulmoBind

INTERVENTIONS:
Drug: PulmoBind — PulmoBind is a peptide derived from human adrenomedullin (hAM1-52), labelled with 99mTc (imaging isotope used in clinical medicine).

SUMMARY:
Pulmonary hypertension or elevation of the pressure in the pulmonary vessels, results from various clinical conditions. It may be idiopathic (of unknown cause) or associated with numerous diseases including cardiovascular and lung disorders. Affected individuals suffer from progressive shortness of breath and, in its most sever forms; pulmonary hypertension carries a worse prognosis than many types of cancer. There is no test currently that can easily and non-invasively detect abnormalities of the pulmonary circulation. Presently there is no cure for pulmonary hypertension and substantial research efforts are dedicated to the development of new drugs that will stop progression or better yet, reverse the disease process. The investigators do not know if any of the drugs currently commercialized for pulmonary hypertension directly improve the status of the pulmonary vessels since no test currently provides this information. Direct earlier detection of lung vessel abnormalities associated with pulmonary hypertension using a sensitive and non-invasive test would allow not only earlier testing of these and of new drugs, but would provide a much better surrogate of disease severity allowing more efficient pre-clinical drug testing. The aim of this phase II study is to evaluate the safety of PulmoBind in participants with pulmonary hypertension and its potential to detect abnormal pulmonary circulation associated within pulmonary hypertension.

DETAILED DESCRIPTION:
Currently there is only one radiopharmaceutical agent approved in Canada (and the world) for clinical imaging of the pulmonary circulation, metastable isotope 99 of technetium. This agent is exclusively used for the diagnosis of physical defects of the circulation due to pulmonary embolus. There is imperative need for new lung tracers that will provide a greater safety profile while enabling functional as well as anatomical imaging of the pulmonary circulation. A novel adrenomedullin derivative has been developed, for molecular imaging of the pulmonary circulation. PulmoBind is labelled with metastable isotope 99 of technetium, the most commonly used imaging isotope in clinical nuclear medicine. PulmoBind is a adrenomedullin derivative specifically designed to bind to the adrenomedullin receptor while avoiding any hemodynamic effects. This novel tracer has the potential to help in the diagnosis and follow-up of various disorders of the pulmonary circulation for which there is currently no alternative. In PulmoBind I three escalating doses were administered and safety was assessed. The product was well tolerated and there were no safety concerns. Imaging revealed predominant lung uptake.

ELIGIBILITY:
HEALTHY VOLUNTEERS:

Inclusion Criteria:

* Male of female participants greater than 18 years of age,
* Female participants must be post-menopausal (defined as two year after last menstrual cycle) or surgically sterilized or use 1 form of contraception with a urine negative pregnancy test (commercial brand: first response kit) within 2 hours of study drug injection,
* Baseline measurements must be within limits of normal or judged non-clinically significant by the investigator:

  * Blood pressure systolic 90 mmHg to 140 mmHg,and diastolic 50 mmHg to 90 mmHg;
  * Heart rate: 50 to 100 beats per minute;
  * Oral temperature: less than 37.6C;
  * Respiratory rate: 12 to 20 breaths per minute;
  * Lung function testing within 6 months;
  * Electrocardiogram in the past three years;
  * Chest X-Ray in the past three years;
  * Electrocardiogram.

Exclusion Criteria:

* Any known chronic or acute medical condition with or without the need for chronic pharmacologic therapy or any condition that may interfere with normal biodistribution of PulmoBind. This includes but is not restricted to: lung parenchymal or lung vascular diseases such as chronic obstructive pulmonary disease, bronchitis, lung cancer, pleural effusion, emphysema, asthma, pulmonary fibrosis, occupational lung disease,pulmonary hypertension (primary or secondary), systemic hypertension, diabetes, cancer, kidney disease, liver disease, heart failure or previous myocardial infarction, coronary artery disease, peripheral vascular disease or inflammatory disease,
* Participants requiring chronic administration of any substance for a medical condition,
* Active smoking or history of smoking within 6 months,
* Alcoholism or known substance abuse,
* Psychotic,addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements,
* Unable to tolerate study procedures (e.g. venipuncture, movement restrictions during imaging),
* Previous nuclear medicine study within one week (to avoid cross-contamination).

PULMONARY HYPERTENSION PARTICIPANTS:

Inclusion Criteria:

* Male of female participants greater than 18 years of age and upper age 70,
* Female participants must be post-menopausal (defined as two year after last menstrual cycle) or surgically sterilized or use 1 form of contraception with a urine negative pregnancy test (commercial brand: first response kit) within 2 hours of study drug injection,
* Diagnosis of pulmonary hypertension (PH) according to the Dana Point PH classification of the following types:

  * Type I: idiopathic, heritable or scleroderma spectrum of disease,
  * Type IV: unoperated chronic thromboembolic PH.
* Participants with chronic thromboembolic pulmonary hypertension (CTEPH) must have a previous positive V/Q scan and multiple chronic/organised occlusive thrombi/emboli in the pulmonary arteries (main, lobar, segmental, subsegmental) on CT angiogram or conventional pulmonary angiography,
* Documented hemodynamic diagnosis of significant PH by right heart catheterization - performed at any time prior to Screening showing:

  * Resting mean pulmonary arterial pressure (mPAP) > 25 mmHg and
  * Resting pulmonary vascular resistance (PVR) > 240 dyn/s.cm5 and
  * Resting capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVDEP) ≤ 15 mmHg (if available),
* New York Heart Association (NYHA) functional class II-III,
* Six minutes walking distance test of ≥ 250 meters, and ≤ 450 meters within 6 months,
* Echocardiogram documented in the participants medical history (including an agitated saline study),
* Computed tomography of the chest documented in the participants medical history.

Exclusion Criteria:

* Participants with impaired renal function defined as estimated creatinine clearance ≤ 30 ml/min (eGFR with modification of diet in renal disease (MDRD) calculator formula),
* Significant liver impairment:

  * Aspartate alanine transferase ( ALT) and/or Aspartate transaminase (AST) ≥ 3 x upper limit of normal (ULN)
  * Bilirubin ≥ 1.5x ULN ( > 35% direct bilirubin)
* Unstable pulmonary arterial hypertension defined as recent syncope or World Health Organization (WHO) functional class IV,
* Participants with CTEPH not on anticoagulant therapy,
* Echocardiographic restrictive lung disease (total lung capacity < 70% of predicted) or obstructive (FEC1/Forced Vital Capacity < 70%),
* Systemic blood pressure < 90 mmHG systolic or less than 50 mmHG diastolic,
* Patient foramen ovale with significant right to left shunting with hypoxia (room air saturation < 88%),
* Active smoking within six months,
* More than minimal pulmonary fibrosis on high resolution computed tomography of the chest,
* The subject's clinical condition is such that they are not expected to remain clinically stable for the duration of the study,
* Active coronary artery disease or stable coronary artery disease that has required an intervention or any change of therapy within 6 months,
* Alcoholism or known substance abuse,
* Psychotic,addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements,
* Participants who have participated in a clinical study involving another investigational drug or devise within four weeks before screening,
* Female participants who are pregnant or breastfeeding,
* Previous nuclear medicine study within one week,
* Unable to tolerate study procedures (e.g. venipuncture, movement restrictions during imaging).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To determine the absence of allergic reaction after repeated exposures to PulmoBind in healthy participants | Static lung uptake 10 minutes duration post injection
To determine the safety of PulmoBind in participants diagnosed with pulmonary hypertension. | Static lung uptake 10 minutes duration post injection
To determine the capacity of PulmoBind lung scan for the detection of abnormal pulmonary circulation associated with pulmonary hypertension. | Status lung uptake 10 minutes duration post injection
  This is an efficacy outcome

SECONDARY OUTCOMES:
To determine the intra-subject variability for quantification of PulmoBind lung uptake in control participants | Status lung uptake 10 minutes duration post injection
Determine the capacity of PulmoBind lung scan to diagnose pulmonary perfusion defects in participants with chronic thromboembolic pulmonary hypertension. | Status lung uptake 10 minutes duration post injection
To correlate lung PulmoBind scan results with parameters of the severity of pulmonary hypertension: 6 minutes walking distance, New York Heart Association functional class, pulmonary artery pressure measured by echo, pulmonary artery pressure measured by | Status lung uptake 10 minutes duration post injection

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Dupuis, MD, Principal Investigator — Montreal Heart Institute
Locations (3):
- Canada (3):
  - Montreal Heart Institute, Montreal, Quebec
  - Sir Mortimer B.Davis Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Harel F, Langleben D, Provencher S, Fournier A, Finnerty V, Nguyen QT, Letourneau M, Levac X, Abikhzer G, Guimond J, Mansour A, Guertin MC, Dupuis J. Molecular imaging of the human pulmonary vascular endothelium in pulmonary hypertension: a phase II safety and proof of principle trial. Eur J Nucl Med Mol Imaging. 2017 Jul;44(7):1136-1144. doi: 10.1007/s00259-017-3655-y. Epub 2017 Feb 24. PMID 28236024